CLINICAL TRIAL: NCT00494793
Title: Vacuum Assisted Wound Closure (VAWC) and Mesh Mediated Fascial Traction - Prospective Study of a Novel Technique for Open Abdomen Closure
Brief Title: Vacuum Assisted Wound Closure (VAWC) and Mesh Mediated Fascial Traction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Collaborators: Uppsala University Hospital (Other); Gävle Hospital (Other); Falu Hospital (Other); KCI Europe Holding B.V. (Industry); The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Ulf Petersson, MD, PhD, Ass prof, Skane University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPNLund 564/2005
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Open Abdomen; Fascial Closure
Keywords: Open abdomen; Fascial closure; Vacuum assisted wound closure; Mesh; Abdominal compartment syndrome; Intraabdominal pressure; Incisional hernia
MeSH Terms: conditions — Intra-Abdominal Hypertension; Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VAWC and mesh mediated fascial traction (Other): This is a study aiming to evaluate one technique for temporary abdominal closure for open abdomen therapy in all patients applicable according to the inclusion criteria
  Interventions: Procedure: VAWC and mesh mediated fascial traction

INTERVENTIONS:
Procedure: VAWC and mesh mediated fascial traction — The first period of 2-5 days only the abdominal VAWC dressing is applied. On day 3-10 a polypropylene mesh is sutured to the fascial edges, between the two layers of the VAWC system, and tightened.
  The VAWC dressing is changed and the mesh tightened every 2-3 days, resulting in gradual approximation of the fascial edges.
  Finally the mesh is removed and the fascia is closed

SUMMARY:
The purpose of this multicenter trial is to prospectively evaluate a novel combination of vacuum assisted wound closure (VAWC) and mesh mediated fascial traction for closure of open abdomens.

DETAILED DESCRIPTION:
Open abdomen treatment often results in difficulties in closing the abdomen. Highest closure rates are seen with the vacuum assisted wound closure (VAWC) technique. Failures with this technique is occasionally experienced, especially in cases with severe visceral swelling needing longer treatment periods with open abdomen. A novel combination of vacuum assisted wound closure and mesh mediated fascial traction for managing the open abdomen was therefore developed and initially tested in a small pilot-like study with encouraging results with late primary closure of the abdomens in all seven patients.

In this multicenter study we prospectively evaluate the technique.

Inclusion criteria:

All patients treated with open abdomen at the 4 participating hospitals are registered, and only those patients who have commenced therapy with VAWC and mesh mediated fascial traction will be included in the study in an intention to treat model.

Exclusion criteria:

Treatment of open abdomen with other techniques.

Method:

* The first period of 2-5 days only the abdominal VAWC dressing is applied.
* On day 3-10 a polypropylene mesh is sutured to the fascial edges, between the two layers of the VAWC system, and tightened.
* The VAWC dressing is changed and the mesh tightened every 2-3 days, resulting in gradual approximation of the fascial edges.
* Finally the mesh is removed and the fascia is closed.
* At closure the wound to suture length is registered.

Primary endpoint:

Frequency of primary fascial closure.

Secondary endpoints:

* study of factors associated with failure of fascial closure and in-hospital mortality,
* abdominal pressure variation attributable to the use of the technique,
* duration of treatment with open abdomen,
* frequency of incisional hernia after one and five years.

Duration of the study:

3-5 years. Enrollment of open abdomen cases.

Follow-up schedule for patients:

* Clinical evaluation at 1 and 5 years.
* CT-examination at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* open abdomen patients with midline incisions, where vacuum assisted wound closure system and mesh mediated fascial traction is applicable

Exclusion Criteria:

* open abdomen patients treated otherwise

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2006-04-01 (Actual); Primary Completion 2009-08-31 (Actual); Study Completion 2015-04-01 (Actual)

PRIMARY OUTCOMES:
Primary fascial closure rate | 2 months
  Primary fascial closure rate with the technique

SECONDARY OUTCOMES:
Factors associated with failure of fascial closure and in-hospital mortality, abdominal pressure, duration of treatment with open abdomen, frequency of incisional hernia development | 5 years
  Early, intermediate and late outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Petersson, MD, PhD, Principal Investigator — Department of Surgery, Malmö University Hospital, Sweden
Locations (5):
- Sweden (5):
  - Department of Surgery, Falu Hospital, Falun
  - Department of Surgery, Gävle Hospital, Gävle
  - Department of Surgery, Malmö University Hospital, Malmo
  - Department of Vascular Surgery, Malmö University Hospital, Malmo
  - Department of Surgery, Uppsala University Hospital, Uppsala

REFERENCES:
- [Derived] Bjarnason T, Montgomery A, Ekberg O, Acosta S, Svensson M, Wanhainen A, Bjorck M, Petersson U. One-year follow-up after open abdomen therapy with vacuum-assisted wound closure and mesh-mediated fascial traction. World J Surg. 2013 Sep;37(9):2031-8. doi: 10.1007/s00268-013-2082-x. PMID 23703638
- [Derived] Sorelius K, Wanhainen A, Acosta S, Svensson M, Djavani-Gidlund K, Bjorck M. Open abdomen treatment after aortic aneurysm repair with vacuum-assisted wound closure and mesh-mediated fascial traction. Eur J Vasc Endovasc Surg. 2013 Jun;45(6):588-94. doi: 10.1016/j.ejvs.2013.01.041. Epub 2013 Mar 1. PMID 23465456